CLINICAL TRIAL: NCT00984399
Title: Serum Estradiol Levels In Postmenopausal Women With Breast Cancer Receiving Adjuvant Aromatase Inhibitors and Vaginal Estrogen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-110
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2024-05

CONDITIONS: Atrophic Vaginitis; Breast Cancer
Keywords: vaginitis; Postmenopausal; 17-β estradiol; 09-110
MeSH Terms: conditions — Atrophic Vaginitis; Breast Neoplasms; Vaginitis | interventions — Estradiol; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- vaginal 17β-estradiol, questionnaire , symptom checklist (Experimental): This is a prospective longitudinal pilot study, and the targeted patient population is postmenopausal women with breast cancer being treated with adjuvant aromatase inhibitors who are initiated on vaginal 17β-estradiol to relieve symptoms of atrophic vaginitis.
  Interventions: Drug: Vagifem® (vaginal 17β-estradiol) questionnaire & menopause symptom checklist

INTERVENTIONS:
Drug: Vagifem® (vaginal 17β-estradiol) questionnaire & menopause symptom checklist — The goal is to have 30 patients on letrozole and 30 on anastrozole who are initiated on vaginal estrogen for symptoms of urogenital atrophy. All subjects will receive 10mcg vaginal 17-β estradiol tablets. Each subject will serve as her own control. We will monitor serum estradiol and follicle stimulating hormone (FSH) levels closely from 0-24 weeks. We will measure serum estradiol and FSH levels at baseline, and subsequently at weeks 2, 7, 12, 18 and 24 after commencing therapy with 10mcg vaginal 17-β estradiol.
  Other Names: The bloodwork will take less than one hour to perform and will be drawn +/- 72hrs from the date the; patient is due for bloodwork.Baseline bloodwork will be drawn within 14 days of study enrollment prior to the initiation of vaginal 25μg 17- β estradiol.; Patients will be encouraged to come for their research bloodwork 12-24 hours after the insertion of the vaginal 25μg 17- β estradiol tablets.; Patients will record in their diary the time of their last vaginal 10μg 17- β estradiol; tablet insertion. Since we do not know the clinical significance of transient; estradiol elevation in these patients, both the patients and the investigators; will be blinded to the results of these assays for the 24 weeks of study; therapy. We will administer the FSFI survey questionnaire and menopause symptom; checklist at baseline, week 12 and week 24.

SUMMARY:
The purpose of this study is to see if Vagifem® 10mcg is safe for women who have had breast cancer. Vagifem is an estrogen product. It is a tiny tablet that is inserted into the vagina. It relieves vaginal dryness. Women who have had breast cancer are usually told not to take estrogen. This is because estrogen use can lead to a breast cancer recurrence or a new primary breast cancer. It is unclear if the estrogen in Vagifem is only absorbed in the vagina. It may be absorbed into the blood stream for a short time and may cause a brief rise in your estrogen level. However, there is no clear evidence that this would cause any bad effects in patients with breast cancer. How much, if any, of these topical estrogens are absorbed through the vagina is not known. We also do not know what the impact is of low dose estrogen absorption on breast cancer outcomes. Also, the absorption should decrease as the mucus membranes are restored after estrogen exposure.

ELIGIBILITY:
Inclusion Criteria:

* History of breast cancer, stages I-III with pathology confirmed at MSKCC
* Women who have completed all of their primary treatment (surgery, radiation therapy, adjuvant chemotherapy) with the exception of endocrine therapy and currently have no clinical evidence of disease.
* Women who are currently on aromatase inhibitors for at least three months--either letrozole or anastrozole
* Women with symptomatic urogenital atrophy: vaginal dryness, irritation, pruritus, dyspareunia, urinary frequency and/or urinary incontinence
* Menopausal at study entry defined as:

  * Bilateral salpingo-oophorectomy independent of age
  * If natural menopause, age ≥ 50 with cessation of menses for at least 12 months
  * If menopause induced by chemotherapy, age ≥ 50 with no menstrual period at least 12 months after chemotherapy finished
* At least 18 years of age
* Able to participate in the informed consent process
* Gynecology examination within six months
* Able to read/speak English

Exclusion Criteria:

* Inability to give informed consent
* Vaginal bleeding of unknown etiology within 12 months of study entry
* History of prior vaginal 17-β estradiol or other topical estrogen use within the past six months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-09-22 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Letrozole; Anastrozole: This is a prospective longitudinal pilot study, and the targeted patient population is postmenopausal women with breast cancer being treated with adjuvant aromatase inhibitors who are initiated on vaginal 17β-estradiol to relieve symptoms of atrophic vaginitis.
Period: Overall Study
Arm/Group | Letrozole | Anastrozole
Started | 12 | 19
Completed | 8 | 14
Not Completed | 4 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Pts did not start treatment | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Anastrozole | Total
Number analyzed (Participants) | 12 | 19 | 31
Age, Continuous [Median (Full Range); unit: years] | 55 [47 to 70] | 56 [46 to 73] | 55 [46 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 31
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 18 | 26
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 18 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Estradiol From Baseline to Week 12
Description: To determine the change in estradiol and follicle stimulating hormone (FSH) from baseline to twelve weeks in postmenopausal women receiving adjuvant aromatase inhibitors during treatment with low dose vaginal 10 µg 17- β estradiol.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 12 | 19
pg/ml
  Baseline estradiol | 5.21 [0.6 to 9.8] | 4.46 [1.3 to 8.8]
  Week 12 estradiol | 5.23 [1 to 8.7] | 6.72 [1.9 to 18]
  Baseline follicle stimulating hormone (FSH) | 70.92 [36.4 to 121.2] | 68.29 [19.9 to 114.5]
  Week 12 follicle stimulating hormone (FSH) | 71.67 [33.6 to 115.9] | 63.28 [23.4 to 90.5]

2. Secondary Outcome: To Compare the Rise in Estradiol in Women on Letrozole vs. Anastrozole During Treatment With Low Dose Vaginal 10 µg 17- β Estradiol to See if There Are Differences Between Aromatase Inhibitors.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 12 | 19
pg/ml
  Baseline Estradiol | 5.21 [0.6 to 9.8] | 4.46 [1.3 to 8.8]
  Week 12 Estradiol | 5.23 [1 to 8.7] | 6.72 [1.9 to 18]

3. Secondary Outcome: Change in Serum Estradiol Baseline to Week 24
Description: To describe patterns of estradiol over the twenty-four week study period.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: pg/ mL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 12 | 19
pg/ mL
  Baseline Estradiol | 5.21 [0.6 to 9.8] | 4.46 [1.3 to 8.8]
  Week 24 Estradiol | 7.55 [3.5 to 21.6] | 9.26 [3.3 to 23.7]

4. Secondary Outcome: Change in FSH Levels Baseline to Week 24
Description: To describe patterns of FSH levels over the twenty-four week study period.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: mIU/ml
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 12 | 19
mIU/ml
  Baseline FSH | 70.93 [36.4 to 121.2] | 9.26 [3.3 to 23.7]
  Week 24 FSH | 74.07 [35.3 to 105.3] | 70.51 [27.9 to 114.9]

5. Secondary Outcome: To Compare the Patient's Female Sexual Function Index (FSFI) Scores and Menopause Quality of Life Questionnaire at Baseline
Description: The FSFI measures six domains of sexual function: desire, arousal, lubrication, orgasm, satisfaction and pain. An increase in FSFI score means better sexual function. The individual domain scores and full scale score of the FSFI are derived by the computational formula outlined in the table below. Individual domain scores are obtained by adding the scores of the individual items that comprise the domain and multiplying the sum by the domain factor (see below). The full scale score is obtained by adding the six domain scores. It should be noted that within the individual domains, a domain score of zero indicates that no sexual activity was reported during the past month.
  Domain Questions Score range Factor Minimum score Maximum score Desire 1, 2 1-5 0.6 1.2 6.0 Arousal 3, 4, 5, 6 0-5 0.3 0 6.0 Lubrication 7, 8, 9, 10 0-5 0.3 0 6.0 Orgasm 11, 12, 13 0-5 0.4 0 6.0 Satisfaction 14, 15, 16 0 (or 1)-5 0.4 0 6.0 Pain 17, 18, 19 0-5 0.4 0 6.0 Full Scale Score Range 2.0 36.0
Time Frame: Baseline
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 12 | 19
units on a scale | 14.61 [2.7 to 26.2] | 16.01 [5.2 to 25.9]

6. Secondary Outcome: To Compare the Patient's Female Sexual Function Index (FSFI) Scores and Menopause Quality of Life Questionnaire at Baseline, Week 12
Description: as for outcome 5
Time Frame: Week 12
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 12 | 19
units on a scale | 17.75 [3 to 29.6] | 18.87 [3 to 29.6]

7. Secondary Outcome: To Compare the Patient's Female Sexual Function Index (FSFI) Scores and Menopause Quality of Life Questionnaire at Baseline, Week 24
Description: The FSFI measures six domains of sexual function: desire, arousal, lubrication, orgasm, satisfaction and pain. The individual domain scores and full scale score of the FSFI are derived by the computational formula outlined in the table below. Individual domain scores are obtained by adding the scores of the individual items that comprise the domain and multiplying the sum by the domain factor (see below). The full scale score is obtained by adding the six domain scores. It should be noted that within the individual domains, a domain score of zero indicates that no sexual activity was reported during the past month.
  Domain Questions Score range Factor Minimum score Maximum score Desire 1, 2 1-5 0.6 1.2 6.0 Arousal 3, 4, 5, 6 0-5 0.3 0 6.0 Lubrication 7, 8, 9, 10 0-5 0.3 0 6.0 Orgasm 11, 12, 13 0-5 0.4 0 6.0 Satisfaction 14, 15, 16 0 (or 1)-5 0.4 0 6.0 Pain 17, 18, 19 0-5 0.4 0 6.0 Full Scale Score Range 2.0 36.0
Time Frame: Week 24
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 12 | 19
units on a scale | 18.32 [2 to 30.8] | 21.09 [5.3 to 30.8]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Letrozole | Anastrozole
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/19
Other Adverse Events (participants affected / at risk) | 0/12 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT00984399/Prot_SAP_000.pdf